CLINICAL TRIAL: NCT05622279
Title: Percutaneous Needle Tenotomy Associated With Platelet-rich Plasma Injection Platelet-rich Plasma in the Treatment of Refractory Plantar Fasciitis: a Pilot Study of the Effect on Pain and Tolerance
Acronym: ANTILOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Regen Lab SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC22_0153
Record Dates: First submitted 2022-11-13; First posted 2022-11-18 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Plantar Fascitis
Keywords: Plantar fasciitis, needle tenotomy, ultrasound, platelet rich plasma
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Intervention Model Description: The VAS pain data will be compared between before the procedure and 6 months after using a Wilcoxon ranks test for paired data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- percutaneous tenotomy + PRP (Experimental): There will be a single arm receiving the treatment being evaluated
  Interventions: Procedure: Percutaneous tenotomy + PRP

INTERVENTIONS:
Procedure: Percutaneous tenotomy + PRP — The patients will receive a percutaneous ultrasound-guided treatment including a needle tenotomy followed by a PRP injection in the plantar fasciitis.

SUMMARY:
There are various treatments for plantar fasciitis, including physical therapy, orthopedic inserts or steroid infiltrations. However, it is estimated that about 20% of patients do not respond to first-line treatment [Rompe, Sports Med Arthrosc Rev, 2009]. It is therefore necessary to be able to integrate new treatments into the management of this condition. The objective of the study is to assess the effect on pain and the safety of the percutaneous ultrasound-guided tenotomy associated with a platelet rich plasma injection to treat refractory plantar fasciitis.

DETAILED DESCRIPTION:
* Pre-inclusion visit (consultation for scheduling the procedure) After verification of the inclusion criteria, the investigating rheumatologist will inform the patient of the study and give him/her the information note. The patient will be offered a period of reflection before signing the consent form. As the procedure requires prior precautions, this will allow the patient to become aware of them. The patient will be given a prescription for a walking boot and a pair of walking sticks.
* Inclusion visit (D0)

After verification of all the inclusion and non-inclusion criteria, the following examinations will be performed during the inclusion visit before the procedure:

* Signature of the consent by the patient and the investigator
* Interrogatory including collection of concomitant treatments, evaluation of the walking perimeter, evaluation of sports activities
* Clinical examination of the foot (Heel tenderness index)
* Standard X-ray of the foot (if not performed at screening)
* Plantar ultrasound = echogenicity of the plantar aponeurosis, measurement of thickness in mm, search for hypervascularization by Doppler
* VAS pain during activity
* FAAM self-questionnaire
* Procedure in 3 steps:

  1. Local anesthesia by tibial block 60 minutes before the tenotomy
  2. Venous sampling of 10 ml and centrifugation for 5 minutes
  3. Needle tenotomy and injection of 1 ml of PRP at the end of the procedure
* Prescription of enoxaparin at a preventive dose for 7 days

The tolerance of the procedure will be evaluated immediately after the procedure, using a VAS for pain. This will be collected by a nurse. We will also collect the acceptability of the procedure as well as the immediate complications (vagal discomfort, bleeding at the injection site).

The patient will then be monitored for two hours (4 times) in order to verify the lifting of the sensory block and the pain during it.

At the end of the consultation, the patient will receive a patient logbook to be completed at home in the 7 days following the procedure and at 14 days (collection of pain at the injection site and possible side effects) and a second logbook to be completed 6 weeks after the procedure.

-First protocol follow-up at home: D7 The patient will have filled out a daily pain VAS and notified any side effects related to the procedure and the analgesic intake during the first week.

A telephone contact will be made at this date by an investigating physician, or a mandated person, in order to ensure that the logbook has been filled out correctly and that there are no complications. The call will also remind the patient to return the questionnaire by mail (stamped and addressed envelope provided).

- Second protocol follow-up at home: S6 +/- 3 days

Six weeks after the procedure, the patient will complete the patient booklet given at D0 at home:

* FAAM self-questionnaire
* VAS pain during activity
* Occurrence of complications
* Gait perimeter
* Third protocol follow-up: consultation at M3 +/- 7 days A follow-up consultation is performed 3 months after the procedure. This corresponds to the usual follow-up of the patient.

During the consultation, the following examinations will be performed

* Clinical examination (HTI)
* Ultrasound of the foot
* VAS pain during activity
* Complications
* FAAM self-questionnaire
* Gait perimeter
* Questions about returning to sport
* Fourth protocol follow-up: consultation at M6 +/- 7 days (main objective) During the consultation, the following examinations will be performed
* Clinical examination (HTI)
* Ultrasound of the foot
* VAS pain during activity
* Complications
* FAAM self-questionnaire
* Gait perimeter
* Questions about returning to sport

ELIGIBILITY:
Inclusion Criteria :

Patient with chronic inferior heel pain diagnosed as plantar fasciitis plantar fasciitis evolving for more than 3 months with a pain VAS at activity ≥ 4/10

* Failure of the initial management including physical therapy, adaptation of footwear and local steroid infiltration
* Patient 18 years of age or older
* Patient affiliated to a social security plan
* Patient able to understand the protocol and having signed an informed informed consent

Exclusion Criteria :

* Patients on NSAIDs and refusing to discontinue them 1 week and 1 week after the procedure
* Corticosteroid infusion at the same lesion site in the last 3 months
* History of PRP injection at the same lesion site
* Treatment with antiplatelet agents [Acetylsalicylic acid (Aspegic, Kardegic, Duoplavin, Resitune, Asasantine), Clopidogrel (Plavix, Duoplavin), Dipyridamole (Persantine, Cleridium, Asasantine)]
* Coagulation disorders: thrombocytopenia < 150,000 platelets/mm3 - Patients on curative anticoagulants
* Any medical condition that may interfere with pain assessment
* Current hematological disease or in remission for less than 5 years (hematological malignancies, myelodysplasia, autoimmune thrombocytopenia), chemotherapy
* Infection at the time of inclusion (bacterial infection and/or presence of fever and/or antibiotic treatment)
* Pregnant or breastfeeding women or those refusing effective contraception
* Patient deprived of liberty or under legal protection (guardianship or curatorship)
* Patients under court protection
* Patients participating in another clinical research protocol involving a drug or medical device
* Patients unable to follow the protocol, as determined by the investigator
* Patient refusing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the evolution of plantar pain after treatment combining needle tenotomy and PRP injection in refractory plantar fasciitis. | 6 months
  VAS pain at activity

SECONDARY OUTCOMES:
Evaluate the tolerance of the procedure | 6 weeks, 3 months, 6 months
  To evaluate the tolerance of the procedure, a VAS [0 to 10] will be filled in by the patient to evaluate the pain felt during the procedure.
Evaluate the acceptability of the procedure | 6 weeks, 3 months, 6 months
  To assess the acceptability of the procedure, the following question will be asked: Would you be willing to repeat this procedure if necessary?
Evaluate the evolution of the functional discomfort | 6 weeks, 3 months, 6 months
  To evaluate the effect on function, we will use two parameters: the FAAM self-questionnaire and the walking perimeter. The FAAM (Foot and Ankle Ability Measure) self-questionnaire will be completed by the patient before the procedure and then 6 weeks, 3 months and 6 months after the procedure. The score is composed of 21 items evaluating the discomfort in daily activities and 8 in sports activities. The walking perimeter (distance the patient can walk without stopping) will be evaluated at 6 weeks, 3 months and 6 months. It will be assessed by the following scale: Unlimited / More than 1 Km / From 500 to 1000m / From 100 to 500m / Less than 100m / Walking impossible.
Evaluate the return to sports activities | 6 weeks, 3 months, 6 months
  To evaluate the return to sport, the following 3 questions will be asked to the patient: Have you resumed your sport activity? If yes, how long after the infiltration? Was it possible to resume the activity at the same level as before? This will be collected at 3 and 6 months.
Evaluate the evolution of pain when pressing the insertion of the plantar fascia | 6 weeks, 3 months, 6 months
  The HTI (physician-assessed Heel Tenderness Index) score will be assessed before the procedure and after 3 and 6 months. It is a score ranging from 0 to 3 (0 = no pain; 1 = pain; 2 = pain and grimace; 3 = pain, grimace, and foot removal).
Evaluate the evolution of the ultrasound data | 6 weeks, 3 months, 6 months
  Two items will be evaluated before the procedure and after 3 and 6 months:
  * Thickness of the superficial plantar fascia at the insertion
  * Doppler hypervascularization

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France, France

IPD SHARING:
Plan to Share IPD: No